CLINICAL TRIAL: NCT02942914
Title: A First-in-Human, Ascending-Dose Study to Investigate the Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of a Single, Subcutaneous Dose of LY3209590
Brief Title: A Study of LY3209590 in Healthy Participants and Participants With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 16129; I8H-MC-BDCA (Other: Eli Lilly and Company); 2016-001048-20 (EudraCT Number)
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- LY3209590 (Experimental): LY3209590 administered subcutaneously (SC).
  Interventions: Drug: LY3209590
- Placebo (Placebo Comparator): Placebo (sterile saline) administered SC.
  Interventions: Drug: Placebo
- Insulin Glargine (Lantus) (Active Comparator): Insulin Glargine administered SC.
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: LY3209590 — Administered SC
  Arms: LY3209590
Drug: Placebo — Administered SC
  Arms: Placebo
Drug: Insulin Glargine — Administered SC
  Arms: Insulin Glargine (Lantus)

SUMMARY:
This trial is conducted to evaluate the safety of a study drug given by injection under the skin to healthy participants and participants with type 2 diabetes. It will also investigate how the body processes the study drug and the effect of the study drug on blood sugar levels. Information about any side effects and tolerability will be documented. This study is approximately 30 days for each participant, not including screening. Screening is required within 28 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

For all study participants:

* Must be a male, or a female who cannot become pregnant, and who is either a healthy participant, or who has type 2 diabetes for at least 1 year
* Male participants with female partners who can become pregnant must agree to use an effective method of birth control during the study and for 4 months after study drug dosing
* Have a body mass index (BMI) of greater than 18.5 kilogram per square meter (kg/m²) and less than or equal to 35 kg/m² at screening
* Have blood pressure, pulse rate, blood and urine laboratory test results acceptable for the study
* Have venous access sufficient to allow blood sampling

For participants with Type 2 Diabetes Mellitus (T2DM):

* Have T2DM controlled with diet and exercise alone or are stable on metformin for at least 30 days
* If taken, prescription medications for medical conditions (e.g.antihypertensive agents, aspirin or lipid lowering agents) are stable for at least 4 weeks
* Have a hemoglobin A1c (HbA1c) greater than or equal to 7.0% and less than or equal to 9.5%

Exclusion Criteria:

For all study participants:

* Are currently participating in another clinical study
* Have a history of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction
* Have or used to have health problems or laboratory test results or electrocardiogram (ECG) readings that, in the opinion of the doctor, could make it unsafe to participate or could interfere with understanding the results of the study
* Have donated blood or have had a loss of 500 milliliters (mL) or more in the last 3 months or have had any blood donation within the last month from screening
* Intend to start any new over-the-counter or prescription medications 7 and 14 days before planned dosing

For participants with T2DM:

* Have taken any glucose-lowering medications, other than metformin, including insulin, in the past 3 months before screening
* Have had more than 1 episode of severe hypoglycemia, within 6 months before entry into the study, or have a history of hypoglycemia unawareness or poor recognition of hypoglycemic symptoms
* Have had a blood transfusion or severe blood loss in the past 3 months, or any blood disorder that could interfere with the understanding of the results of the study
* Have received chronic (lasting greater than 14 consecutive days) systemic glucocorticoid therapy (excluding topical, intra-articular, and inhaled preparations) in the 3 past months, or have received any glucocorticoid therapy within 30 days before screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2017-10-18 (Actual); Study Completion 2017-10-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Day 31

SECONDARY OUTCOMES:
Pharmacokinetics: Area Under The Concentration Curve Zero to Infinity (AUC[0-∞]) of LY3209590 | Baseline through Day 31
Pharmacodynamics: Average Glucose from 8-Point Glucose Profiles in Participants with T2DM treated with Placebo or LY3209590 | Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Neuss, Germany